CLINICAL TRIAL: NCT03294707
Title: A Phase 1 Randomized, Placebo-controlled, Single and Multiple Ascending Dose Study of the Tolerability, Pharmacokinetics and Pharmacodynamics of AG10 in Healthy Subjects
Brief Title: Single and Multiple Ascending Dose Study Assessing the Safety, Tolerability, PK and PD of AG10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG10-001
Record Dates: First submitted 2017-09-18; First posted 2017-09-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2018-05

CONDITIONS: Amyloid Cardiomyopathy, Transthyretin-Related
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized with an overall ratio of 3:1 to AG10: placebo within each cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AG10 single oral dose (Experimental): AG10 oral tablet, administered by mouth, once
  Interventions: Drug: AG10 oral tablet
- Placebo single oral dose (Placebo Comparator): Placebo Oral Tablet, administered by mouth, once
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: AG10 oral tablet — Active single ascending dose
  Other Names: Eidos Therapeutics AG10
  Arms: AG10 single oral dose
Drug: Placebo Oral Tablet — Placebo single dose
  Other Names: Matching placebo
  Arms: Placebo single oral dose

SUMMARY:
This is a single center, prospective, randomized, placebo-controlled study of AG10 in healthy adult subjects

DETAILED DESCRIPTION:
Up to 48 healthy volunteers will be given a single dose of AG10 or placebo and be monitored for safety and tolerability over a 5-day period. Up to 48 healthy volunteers will be given multiple doses of AG10 or placebo and be monitored for safety and tolerability over a 15-day period.

ELIGIBILITY:
Inclusion Criteria:

* Weight between >50 kg and ≤110 kg;
* BMI of 18 to 32 kg/m2;
* Subjects who are healthy as determined by medical history, physical examination, 12 lead ECG and standard laboratory tests;
* Subjects who are negative for drugs of abuse and alcohol tests;
* Subjects who are non-smokers;

Exclusion Criteria:

* Subjects who have used prescription drugs within 4 weeks of first dosing;
* Subjects who have a prior cholecystectomy;
* Subjects who have used any over-the-counter medications within 7 days prior to Day -1;
* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders;
* Subjects who have an abnormal screening ECG;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability: individual and summary blood pressures, heart rate, ECG and lab data presented in tabular form with descriptive statistics. Adverse events will be tabulated and summarized by Part A (SAD) vs. B (MAD), and treatment. | 30 days
  To evaluate the safety and tolerability of single and multiple doses of AG10 administered to healthy adult subjects

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: T1/2 | 30 days
  Plasma half-life (t1/2)
Pharmacokinetic Assessments: Tmax | 30 days
  Time to maximum concentration (Tmax)
Pharmacokinetic Assessments: Cmax | 30 days
  Maximum concentration (Cmax)
Pharmacokinetic Assessments: Cmin | 30 days
  Cmin
Pharmacokinetic Assessments: AUC | 30 days
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetic Assessments: Clearance | 30 days
  Apparent clearance (CL/F)
Pharmacokinetic Assessments: volume of distribution | 30 days
  Apparent volume of distribution (Vss/F)
Pharmacodynamic Assessments: Assessments of TTR stabilization will be listed and summarized by part, treatment, and time point using appropriate descriptive statistics. | 30 days
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays, including Fluorescent Polarization Exclusion Assay (FPE) and Immunoblotting (Western Blot) and quantitation of prealbumin (TTR).
Pharmacodynamic Assessments: Western blot | 30 days
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays: Immunoblotting (Western Blot)
Pharmacodynamic Assessments: prealbumin | 30 days
  AG10 binding to and/or stabilization of TTR will be evaluated by established ex vivo assays: quantitation of prealbumin (TTR).
Food effect: AUC | 30 days
  To evaluate the effect of food on the PK of AG10. The log transformed values of total AUC will be analyzed using a linear mixed effect model with formulation, period, sequence, and carryover as fixed effects and subject as a random effect.
Food effect: Cmax | 30 days
  To evaluate the effect of food on the PK of AG10. The log transformed values of Cmax will be analyzed using a linear mixed effect model with formulation, period, sequence, and carryover as fixed effects and subject as a random effect.

CONTACTS AND LOCATIONS:
Overall Officials: Terry O'Reilly, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No